CLINICAL TRIAL: NCT04564157
Title: A Phase III Clinical Trial of Adjuvant Chemotherapy vs Chemoimmunotherapy for Stage IB-IIIA Completely Resected Non-small Cell Lung Cancer (NSCLC) Patients.
Brief Title: New Adjuvant Trial of Chemotherapy vs Chemo-immunotherapy
Acronym: NADIM-ADJUVANT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECP 20/05_NADIM-ADJUVANT; 2020-002088-71 (EudraCT Number)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer; Adjuvant Chemotherapy
Keywords: Lung Diseases; Carcinoma, Non-Small-Cell Lung; Stage IB-IIIA lung cancer; Adjuvant treatment; Carcinoma, Bronchogenic; Immunotherapy; Paclitaxel; Carboplatin; Nivolumab; Immune response; Thoracic Neoplasms; Respiratory Tract Neoplasms; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Diseases; Carcinoma, Bronchogenic; Thoracic Neoplasms; Respiratory Tract Neoplasms | interventions — Carboplatin; Paclitaxel; Nivolumab

STUDY DESIGN:
Intervention Model Description: Design: Open-label, randomised, two arm, phase III, multicentre clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant treatment + Adjuvant maintenance treatment (Experimental): Adjuvant treatment:
  * Paclitaxel: 200mg/m2 infusion over 3 hours
  * Carboplatin: AUC5 at the end of the Paclitaxel infusion
  * Nivolumab: 360 mg intravenous Q3W
  It has to start within 3-10 weeks from surgery and the first administration has to be done within 1-3 days from randomization. 4 cycles will be administered at 21day intervals (QW3) after surgery. A CT-SAN must be done after the 4 cycles of adjuvant treatment. Patients must discontinue treatment if there is evidence of disease relapse.
  After the 4 cycles of chemo-immunotherapy the patient will receive:
  Adjuvant maintenance treatment: Nivolumab: 480 mg IV Q4W It will start after 4 weeks from day 1 cycle 4 of adjuvant treatment. 6 cycles will be administered every 28 days. A CT-SAN must be done within +/- 7 days from day 28 of the 3rd cycle of adjuvant maintenance treatment and within +/- 7 days at the end of the 6th cycle. Patients must discontinue treatment if there is evidence of disease relapse at 3rd cycle CT-SCAN.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Nivolumab
- Control arm: Adjuvant treatment (Active Comparator): Adjuvant treatment:
  * Paclitaxel: 200mg/m2 infusion over 3 hours
  * Carboplatin: AUC5 at the end of the Paclitaxel infusion Adjuvant treatment has to start within 3-10 weeks from surgery and the first administration and has to be done within 1-3 days from randomization. 4 cycles will be administered at 21-day (+/- 3 days) intervals (QW3) after surgery. A CT-SAN must be done after the 4 cycles of adjuvant treatment.
  Observation: 2 observation visits will be done at 3 months and at 6 months from day 21 of cycle 4 of adjuvant treatment.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Structure: The cis-diamino (cyclobutan-1, 1 dicarboxilate) plating. Stability: 24 hours at ambient temperature in 5% glucose, glucosaline or physiologic saline. It is recommended not to dilute with chlorinated solutions for this could affect the carboplatin.
  Route of administration: Intravenous infusion.
  Guidelines of Carboplatin administration: According to the standard of each center.
  Other Names: Paraplatin
Drug: Paclitaxel — Structure: A diterpene whose composition is: 5b, 20-epoxy-1, 2a, 4,7b, 10b, 13a-hexa-hidroxytax-11-en 9 one 4,10-diacetate 2-benzoate 13-ester with (2R,3S)- N-benzoyl-3-phenylisoserine.
  Stability: Concentrations of 0.3-1.2 mg/ml in 5% dextrose or normal saline have demonstrated chemical and physical stability for more that 27 hours at ambient temperature (25ºC approximately). The intact vial must be stored between 15º and 25ºC.
  Guidelines on Paclitaxel administration: Paclitaxel must be administered by infusion over 3 hours in dextrose (D5W) or normal saline (NS). The concentration must not exceed 1.2 mg/ml.
  Other Names: Taxol
Drug: Nivolumab — Structure: Nivolumab is a soluble protein consisting of 4 polypeptide chains.
  Route of administration: Intravenous infusion.
  Product Description: Nivolumab (BMS-936558-01) Injection drug product is a sterile, non-pyrogenic, single-use, isotonic aqueous solution formulated in 10 mg/ml.
  Storage Conditions: It must be stored at 2 to 8 degrees Cº and protected from light and freezing.
  Guidelines: The administration of nivolumab infusion must be completed within 24 hours of preparation.The dose of Nivolumab for the adjuvant treatment is 360 mg administered as an intravenous infusion over 30 minutes every 3 weeks (+/-3 days) for 4 cycles.
  For the maintenance adjuvant treatment the dose is nivolumab 480 mg Q4W (+/-3 days) over 30 minutes for 6 months (6 cycles).
  Subjects should be carefully monitored during nivolumab administration to follow infusion reactions.
  Doses of nivolumab may be interrupted, delayed, or discontinued depending on how well the subject tolerates the treatment.
  Other Names: Opdivo
  Arms: Adjuvant treatment + Adjuvant maintenance treatment

SUMMARY:
This is an open-label, randomised, two-arm, phase III, multi-centre clinical trial.

210 stage IB-IIIA, completely resected, non-small cell lung cancer patients will be enrolled in this trial to evaluate the disease free survival between experimental arm (Adjuvant Chemotherapy-Immunotherapy + maintenance adjuvant Immunotherapy) and control arm (Adjuvant Chemotherapy)

DETAILED DESCRIPTION:
This is an open-label, randomised, two-arm, phase III, multicentre clinical trial.The total sample size is 210 and 105 per arm. The population to be included are stage IB-IIIA, completely resected, non-small cell lung cancer patients.

Patients randomised to the experimental arm will receive Nivolumab 360mg + Paclitaxel 200mg/m2 + Carboplatin AUC5 for 4 cycles every 21 days (+/- 3 days) as adjuvant treatment followed by maintenance adjuvant treatment for 6 cycles with Nivolumab 480 mg Q4W (+/- 3 days).

Patients randomized to the control arm will receive Paclitaxel 200mg/m2 + Carboplatin AUC5 for 4 cycles every 21 days (+/- 3 days) followed by 2 observation visits.

The primary objective is to evaluate the disease-free survival (DFS): defined as the length of time from randomization to the earliest event defined as disease recurrence, any new lung cancer (even in the opposite lung), or death from any cause at any known point in time.

Patient accrual is expected to be completed within 3.5 years, excluding a run-in-period of 3 months. Treatment and follow-up are expected to extend the study duration to a total of 8.5 years. Patients will be followed 5 years after adjuvant treatment or observation phase. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed of primary non-small cell lung cancer, histologically confirmed
* 2. Patients should be classified postoperatively in stage IB (=4 cm), II or IIIA according to pathological criteria and according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology.
* 3. Complete surgical resection of the primary NSCLC is also essential. Surgeons are strongly advised to dissect or obtain samples of all accessible lymph node levels, as established in the European Society of Thoracic Surgeons guide . Consequently, at the end of the surgical intervention it is recommended to have obtained samples of a minimum of 3 (three) specific mediastinal ganglionic lobe stations (N2), one of which should include station 7, and at least one N1 station (including those resected with the tumor piece).
* 4. The surgical intervention may consist of a lobectomy, sleeve resection, bilobectomy or pneumonectomy, as determined by the responsible surgeon based on intraoperative findings. Patients who have had only segmentectomies or wedge resections are not considered eligible for participation in this study.
* 5. Preoperative (neoadjuvant) use of platinum-based chemotherapy or other types of chemotherapy are not accepted.
* 6. Preoperative, postoperative, or scheduled radiation therapy is not accepted for a later time. Patients with only N2 disease, who have to receive post-operative adjuvant radiotherapy will not be eligible.
* 7. A minimum of 3 weeks must have elapsed between the surgical intervention performed for the NSCLC and the randomization. Adjuvant treatment must start between the 3rd and the 10th week from surgery.
* 8. ECOG 0-1
* 9. Patients aged ≥ 18 years
* 10. Correct hematological, hepatic and renal function i. Neutrophils ≥ 1500×109/L ii. Platelets ≥ 100 ×109/L iii. Hemoglobin > 9.0 g/dL iv. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault).v. AST/ALT ≤ 3 x ULN vi. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 x ULN) vii. The patients need to have a forced expiratory volume (FEV1) ≥ 1.2 liters or >40% predicted value viii. INR/APTT within normal limits.
* 11. Patient consent must be obtained in the appropriate manner as established in the applicable local and regulatory requirements
* 12. Patients must be accessible for treatment and follow-up
* 13. Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 3 days before randomization.
* 14. All sexually active men and women of childbearing potential must use a highly effective contraceptive method (two barrier methods or a barrier method plus a hormonal method) during the study treatment and for a period of at least 5 months for females and 7 months for males following the last administration of trial drugs.

Exclusion Criteria:

* 1. Patients with a history of other malignant diseases, with the exception of the following:

  * or properly treated non-melanotic skin cancer
  * or cancer in situ treated with curative intent
  * or other malignancies treated with curative intent and without signs of disease for a period of> 3 years after the end of the treatment and which, in the opinion of the doctor in charge of their treatment, do not present a substantial risk of relapse of the previous malignant disease.
* 2. Patients with ALK, STKB11 o KEAP1 known mutations before inclusion in this trial.
* 3. Patients with adenocarcinoma NSCLC must be tested for the common EGFR mutations before inclusion. Patients with any known EGFR mutation cannot be enrolled in the study.
* 4. Patients with a combination of microcytic and non-small cell lung cancer, a carcinoid lung tumor or large cell neuroendocrine carcinoma.
* 5. Patients that received live attenuated vaccines within 30 days prior to randomization.
* 6. History of a primary immunodeficiency, history of organ allogeneic transplantation, use of immunosuppressive drugs within 28 days before randomization or previous history of toxicity of severe immune mechanism (grade 3 or 4) with other immunological treatments
* 7. Patients with active or uncontrolled infections or with serious medical conditions or disorders that may not allow patient management as established in the protocol
* 8. Patients who have suffered untreated and / or uncontrolled cardiovascular disorders and / or who have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction in the previous year or ventricular cardiac arrhythmias that require medication, history of atrioventricular conduction of second or third degree). Patients with relevant cardiac history, even when well controlled, should have an LVEF> 50% in the 12 weeks prior to randomization
* 9. Pregnant or breastfeeding women
* 10. Patients in whom R0 resection cannot be confirmed
* 11. Patients with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* 12. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* 13. Any positive test result for hepatitis B virus or hepatitis C virus, indicating presence of virus, e.g. Hepatitis B surface antigen (HBsAg, Australia antigen) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative)
* 14. History of allergy or hypersensitivity to any of the study drug components
* 15. Prior anti-PD1/L1 treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
The disease-free survival | From the date of randomization to the date of last follow up, assessed up to 60 months
  The length of time from randomization to the earliest event defined as disease recurrence, any new lung cancer (even in the opposite lung), or death from any cause at any known point in time.

SECONDARY OUTCOMES:
Overall survival | From the date of randomization until the date of last follow up, assessed up to 60 months
  Defined as the time between the date of randomization and the date of death
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From the subject's written consent to participate in the study through 100 days after the final administration of the drug
  It will be measured by the incidence of AE, SAE, immune-related AEs, deaths, and laboratory abnormalities. Adverse events will be graded according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — Fundación GECP President
Locations (30):
- Spain (30):
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Parc Taulí, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital San Pedro De Alcántara, Cáceres
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - ICO Girona, Hospital Josep Trueta, Girona
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Fundación de Alcorcón, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Nuestra Señora La Candelaria, Santa Cruz de Tenerife
  - Hospital Virgen del Rocío, Seville
  - Instituto Valenciano De Oncología, Valencia
  - Hospital Clínico de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Complexo Hospitalario Universitario De Vigo, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org